CLINICAL TRIAL: NCT01627275
Title: Naive T-Cell Depleted Donor Lymphocyte Infusion Following Allogeneic Stem Cell Transplantation
Brief Title: Naive T-Cell Depleted DLI Following Allo Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mitchell Horwitz, MD (Other)
Responsible Party: Sponsor-Investigator, Mitchell Horwitz, MD, Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003975
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Hematological Malignancies
Keywords: Naive T Cell Depletion; Donor Lymphocyte Infusion; Allogeneic Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DLI from HLA-identical donor (Experimental): Naive T Cell Depleted Donor Lymphocyte Infusion from HLA matched family member donor or 8/8 HLA matched unrelated donor.
  Interventions: Biological: Naive T Cell Depleted Donor Lymphocyte Infusion

INTERVENTIONS:
Biological: Naive T Cell Depleted Donor Lymphocyte Infusion — A single naive T-cell depleted donor lymphocyte infusion will be administered through a peripheral or central venous catheter greater than or equal to 60 days post allogeneic hematopoietic stem cell transplant.
  Other Names: CD45RA+ T Cells

SUMMARY:
Allogeneic stem cell transplantation offers the hope of cure for a wide variety of hematologic malignancies. Mature donor T-cells play a critical role in the success or failure of this procedure and a subset of donor T-cells mediate graft-versus-host disease while other subsets provide the foundation for immune recovery. The major challenge in allogeneic stem cell transplantation is determining how to maximally exploit the beneficial effects mediated by T-cells without causing GvHD. This challenge could be overcome by selectively depleting the population of donor T-cells responsible for eliciting the GvHD response. The study hypothesis is depletion of naïve T-cells from the donor lymphocyte inoculum will not cause GVHD while providing T-cells to affect both anti-infection and anti-tumor responses.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation (SCT) offers the hope of cure for a wide variety of hematologic malignancies. Mature donor T-cells play a critical role in the success or failure of this procedure. A subset of donor T-cells mediates graft-versus-host disease (GvHD). Other subsets provide the foundation for immune recovery. Pan-depletion of mature donor T-cells is an obligate step in haploidentical allogeneic stem cell transplantation. Without this step, the recipient would succumb to lethal acute GVHD. We have had extensive experience with in-vivo donor (and recipient) T-cell depletion using alemtuzumab as part of the bone marrow conditioning regimen. We and others have also used anti-thymocyte globulin for the same purpose. Pan-depletion of T-cells eliminates GvHD but significantly increases the risks of tumor relapse and opportunistic infections. A delayed donor lymphocyte infusion augments immune recovery and the graft versus tumor response, but it comes at the risk of inducing lethal GvHD. This is particularly problematic when the donor and recipient are HLA-discordant. Thus the major challenge in allogeneic stem cell transplantation is determining how to maximally exploit the beneficial effects mediated by T-cells without causing GvHD. This challenge could be overcome by selectively depleting the population of donor T-cells responsible for eliciting the GvHD response. We have been interested in selecting T-cells based on their naïve or memory phenotype to understand the contribution of each of these cells to the pathogenesis of GvHD. Naïve T-cells (CD62L+ or CD45RA+) are T-cells that have not encountered antigens specific for their T-cell receptor. Memory T-cells (CD62L- or CD62L+ or CD45RA-) are T-cells that have previously been exposed to their corresponding cognate antigens. If a donor has not encountered host alloantigens, GvHD-inducing host-reactive T-cells should be contained in the naïve T-cell compartment. In contrast, all the memory phenotype cells should not recognize host alloantigens. If this hypothesis is correct as suggested by several published studies, CD62L- T-cells, which are devoid of naïve T-cells and represent a subset of memory T-cells, should not be able to induce GvHD. The study hypothesis is depletion of naïve T-cells from the donor lymphocyte inoculum will abrogate GVHD while providing immunocompetent memory T-cells to affect an anti-infection and a graft versus tumor response. In this study, we will determine the maximum tolerated dose of a naïve T-cell depleted donor lymphocyte infusion given to patients following HLA-matched allogeneic stem cell transplantation. We will assess the GVHD-inducing potential of this donor lymphocyte infusion and further monitor the impact that this DLI will have on post-transplant immune recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone an alemtuzumab or thymoglobulin-containing allogeneic transplant procedure from an HLA-identical family donor, or an 8/8 HLA-matched unrelated donor.
* At least 60 days from day of transplantation.
* Karnofsky performance status 50-100%.
* Donor myeloid engraftment (from peripheral blood or bone marrow) of at least 40% documented ≤ 60 days from protocol therapy.
* No active acute GvHD ≥ grade II.
* Prednisone (or equivalent corticosteroid) dose ≤ 20mg, daily mycophenolate mofetil dose ≤2000mg/d and cyclosporine/tacrolimus at ≤ therapeutic blood trough levels.
* No change in dosing of immunosuppressive agents 2 weeks before the naïve T-cell depleted donor lymphocyte infusion.
* A commitment not to electively taper for a minimum of 60 days, the immunosuppressive medications ongoing at time of naïve T-cell depleted donor lymphocyte infusion.
* No extensive chronic GvHD.
* Age ≥ 18 years of age.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with other major medical or psychiatric illnesses, which the treating physician feels, could seriously compromise tolerance to this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-06; Primary Completion 2017-02-24 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
MTD of Naive TCD DLI | 12 months
  To determine the maximum tolerated dose (MTD) of a Naive T cell depleted (TCD) donor lymphocyte infusion (DLI) post alemtuzumab-containing allogeneic transplant procedure from a HLA-identical family donor, or an 8/8 HLA-matched unrelated donor and derive a preliminary assessment of the efficacy of the naive T-cell depleted DLI.

SECONDARY OUTCOMES:
Immunological Recovery | 12 months
  Immunological recovery will be assessed by the immune function panel which consists of a standardized panel of T-cell, B-cell, NK-cell, and dendritic cell antibodies, measurement of T-cell function, analysis of B-cell recovery, quantification of Naive T-cell recovery and a T-cell repertoire assay.
Overall Incidence of Acute GVHD | 60 Days
  To assess the overall incidence of Acute Graft Versus Host Disease
Overall Incidence of Opportunistic Infections | 60 Days
  To assess the overall incidence of opportunistic infections
Overall Incidence of Chronic GVHD | 12 months
  To assess overall incidence of Chronic Graft Versus Host Disease

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Horwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States